CLINICAL TRIAL: NCT06194669
Title: Mechanisms of Somatic Mutation and Tumor Initiation in Pre-malignant Kidney Tubule Cells
Acronym: SoMuKT
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Irene Franco, Doctor, IRCCS San Raffaele
Other Study IDs: SoMuKT
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Renal Cell; Von Hippel-Lindau Disease
Keywords: Somatic mutations; Whole genome sequencing; Normal kidney
MeSH Terms: conditions — Carcinoma, Renal Cell; von Hippel-Lindau Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine samples, kidney tumor biopsies, kidney cyst biopsies, normal kidney tissue adjacent to tumor biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Healthy volunteers; patients referring to San Raffaele Hospital for renal/urological conditions other than VHL
  Interventions: Other: Blood and urine sample collection
- VHL-disease patients: Individuals with genetic diagnosis of Von Hippel Lindau disease
  Interventions: Other: Blood and urine sample collection

INTERVENTIONS:
Other: Blood and urine sample collection — One whole blood sample per individual (3 ml) will be collected. Up to 5 urine samples per individual will be collected

SUMMARY:
The goal of this observational study is to analyze somatic mutations in the genome of normal kidney cells from patients affected by kidney cancer predisposition syndrome Von Hippel Lindau (VHL) and compare the mutation rates observed in these patients and in individuals not affected by the disease. The main questions the study aims to answer are:

* Do kidney cells from VHL patients mutate more than cells from control individuals during adult life?
* What mechanisms favor somatic mutation occurrence in the genome of normal kidney tubule cells?

Participants will donate one blood sample and multiple urine samples. Urines will be used for kidney cell isolation, followed by cell culturing and genetic analyses. Urine samples will be collected once a year for 3-5 years. Sample collection will occur during the yearly screening program that each patient undergoes at the hospital. In case patients undergo surgical treatment of kidney tumors, samples discarded from surgery (tumor and normal kidney adjacent to tumor) will be collected and subjected to genetic analyses.

Researchers will compare the number and types of mutations found in tumors and normal kidney cells from VHL-disease patients with those found in normal kidney cells from control individuals, to see if somatic mutation rates are increased in VHL-disease patients during aging.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of VHL-disease; age (data need to be collected from a population distributed between 25 and 65 years); gender (males and females should be equally represented);

Exclusion Criteria:

* patients with bilateral nephrectomy, in dialysis or kidney transplant; use of nephrotoxic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with genetic diagnosis of VHL-disease, between 25 and 65, both genders
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of somatic mutation accumulation in normal kidney tubule genomes | Normal kidney tubule cells from urines are assessed from control and VHL-disease patients typically over a period of 3 years (min 3 months, max 3 years)
  The genome of multiple normal kidney cells from each subject will be investigated by whole genome sequencing. The number of somatic mutations per genome will be plotted according to donor's age and a curve describing the accumulation of mutations with age will be obtained for both the control and VHL-disease patient populations. The aim is to assess differences in mutation rates in the kidney of VHL-disease patients vs controls and understand the underlying mechanism.

SECONDARY OUTCOMES:
Quantification of pre-cancer cells in urines | Normal kidney tubule cells from urines are assessed from control and VHL-disease patients typically over a period of 3 years (min 3 months, max 3 years)
  From each urine sample, researchers can culture up to 20 single cell clones and perform a single-clone, gene-expression analysis. The expression of markers that characterize the mutation-prone, pre-cancer population will be assessed in all clones. The fraction of clones expressing markers of pre-cancer cells will be calculated in control and VHL-disease groups. The aim is to assess any differences in the presence of pre-cancer cells in urines from VHL-disease patients vs controls and assess any correlation of this parameter with kidney cancer occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Franco, PhD, Principal Investigator — IRCCS Ospedale San Raffaele; Alessandro Larcher, MD, Principal Investigator — IRCCS Ospedale San Raffaele; Andrea Salonia, MD, Study Chair — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy